CLINICAL TRIAL: NCT07124247
Title: Implementation of the MOX Activity Monitor in Hospitalized Geriatric Rehabilitation
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: KU Leuven (Other)
Collaborators: Universitaire Ziekenhuizen KU Leuven (Other)
Responsible Party: Principal Investigator, Margaretha van Dijk, Principal Investigator, KU Leuven
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: S70120
Record Dates: First submitted 2025-07-25; First posted 2025-08-15 (Actual); Last update posted 2025-08-15 (Actual); Status verified 2025-08

CONDITIONS: Hip Fracture; Stroke; Fraility
Keywords: geriatric patients; geriatric rehabilitation; physiotherapy; activity monitor
MeSH Terms: conditions — Hip Fractures; Stroke

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Patient (Experimental): The participants will be equipped with the MOX activity monitor for one week.
  Interventions: Device: Activity registration for one week with an activity monitor (MOX1)

INTERVENTIONS:
Device: Activity registration for one week with an activity monitor (MOX1) — The participants will be equipped with the MOX activity monitor, which will be attached to the thigh. The device is waterproof, allowing participants to shower and swim, and does not require recharging during the study period.
  The MOX will be attached on the same day as the BBS and Handgrip strength measurements, which will take place on a Friday. The following Monday, the 10mWT will be conducted, thus within the same week that the MOX is attached.
  The MOX monitor will be worn for one week.

SUMMARY:
Staying active is essential for healthy aging, but hospitalized older adults in rehabilitation often move very little. This study explores how much physical activity these patients actually get and how it relates to their recovery. Using the MOX activity monitor-a device that accurately tracks walking, standing, and sedentary time-the study aims to better understand daily activity patterns during rehabilitation.

Researchers will test the best way to use the MOX monitor, develop a standard protocol for its use, and integrate its data into patients' electronic health records. By comparing MOX activity data with standard measures of physical performance, the study will determine how useful activity monitoring is for tracking recovery in older patients. This could lead to improved care and more personalized rehabilitation plans in the future.

DETAILED DESCRIPTION:
Prolonged sitting is a growing public health concern. Adults now spend up to 85% of their day sedentary, and older adults are the most inactive group. Research shows that the negative health effects of prolonged sitting persist even in individuals who engage in regular physical activity. Excessive sedentary behavior is associated with loss of independence, cardiovascular issues, and reduced mental well-being. Recommendations from public health institutions suggest minimizing uninterrupted sitting to no longer than 30 minutes.

In hospitalized geriatric patients, particularly during the acute phase of illness, physical activity often drops drastically. This sudden decline in movement can lead to rapid deconditioning, muscle loss, and reduced ability to perform basic daily activities. As a result, these patients face longer hospital stays and a higher risk of admission to long-term care facilities.

Despite widespread recognition of the importance of daily activity for healthy aging, promoting and monitoring movement in the hospital environment remains a challenge. One key question remains: how active are geriatric rehabilitation patients during their hospital stay?

A previous study (S64932) validated the MOX activity monitor as a reliable tool for measuring daily activity-including time spent walking, standing, and sitting-in hospitalized older adults. However, several important questions remain unanswered:

What is the most effective and reliable way to use the MOX monitor in clinical practice?

How do daily activity levels relate to functional recovery during rehabilitation?

Can advanced parameters from the monitor, such as the number and intensity of sit-to-stand transitions or stair-climbing activity, offer additional insight into lower-limb function?

This study aims to fill these gaps by developing a standardized protocol for implementing the MOX monitor in geriatric rehabilitation wards. It also aims to integrate activity monitor data into existing electronic health systems, including the Interprofessional Dossier (IPD) within the Clinical Work System (KWS). The reliability and usability of this integration will be assessed.

Furthermore, the study will explore the validity of an open-source algorithm-previously validated in community-dwelling older adults-for detecting sit-to-stand transitions in hospitalized geriatric patients. By correlating MOX-derived activity data with established functional outcome measures, the study seeks to determine the clinical value of activity monitoring in rehabilitation settings.

Ultimately, this research supports the functional integration of innovative activity monitoring tools into standard geriatric care, with the goal of improving patient outcomes through better understanding and promotion of physical activity during hospitalization.

ELIGIBILITY:
Inclusion Criteria:

* Hospitalized on the geriatric rehabilitation ward of UZ Leuven, campus Pellenberg
* 70 years or older
* Signed informed consent

Exclusion Criteria:

* Cognitive impairment making it impossible to understand instructions
* Unable to perform the standard of care physical tests 10mWT, BBS, and handgrip

Min Age: 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2025-08-08 (Estimated); Primary Completion 2026-03-01 (Estimated); Study Completion 2026-07-01 (Estimated)

PRIMARY OUTCOMES:
Total minutes of active behaviour (walking/ standing) during one day | 1 year
  Total minutes active (walking and/or standing) during the day, measured with the MOX activity monitor

SECONDARY OUTCOMES:
Number of bouts of sedentary behaviour during a day | 1 year
  Number of bouts of sedentary behaviour during a day., measured with the MOX activity monitor.
Number of free-living sit-to-stand transitions during a day | 2 year
  Validate an open access algorithm of the MOX activity monitor data, to detect and quantify free-living sit-to-stand transitions , in hospitalized geriatric patients requires further investigation. in a sample of hospitalized geriatric patients ( including retrospectively analysing previous data of study S64932).
Number of stair-climbing activity during a day | 2 years
  Detect stair-climbing activity of the MOX activity monitor data, in a sample of hospitalized geriatric patients ( including retrospectively analysing previous data of study S64932).
Functional balance | 2 years
  Functional balance measured with the Berg balane scale
Comfortable walking speed | 1 year
  Comfortable walking speed measures with the10m Walk Test.
Handgrip strength | 1 year
  Handgripstrength measured with the Martin Vigorimeter

CONTACTS AND LOCATIONS:
Locations (1):
- UZ Leuven, campus Pellenberg, Pellenberg, Belgium

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] van Dijk M, Bijnens W, Van Driessche C, Van Meerbeek T, Allegaert P, Van Cleynenbreugel H, Verschueren S, Verheyden G, Tournoy J, Flamaing J. Accuracy of an Activity Monitor in Assessing Physical Activity of Hospitalized Geriatric Rehabilitation Patients With Slow Walking Speed Using a Walking Aid. J Aging Phys Act. 2024 Nov 20;33(3):243-250. doi: 10.1123/japa.2023-0319. Print 2025 Jun 1. PMID 39566489